CLINICAL TRIAL: NCT01889030
Title: Cardiovascular Risk Stratification of Ambulatory Patients in Primary Prevention. RISK Study
Brief Title: Cardiovascular Risk Stratification of Ambulatory Patients in Primary Prevention
Acronym: RISK
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CAR-XXX-2013/1
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Primary Prevention
Keywords: Cardiovascular primary prevention; Cardiovascular risk strtification

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Target population: This observational, cross-sectional, national multicenter designed study will describe the frequency of use of different evaluation methods (risk scores or subjective assessment) employed to determine the cardiovascular risk of patients in a primary care setting, at both General Practitioners (GPs) or Cardiologists offices.

SUMMARY:
This is an observational, cross-sectional, national multicenter study, trying to obtain local data about the global cardiovascular risk profile of patients attending ambulatory offices of general practitioners and cardiologists.

The aim of the study is to describe how physicians diagnose and stratify their patients in cardiovascular primary prevention setting and to highlight if patients are stratify through objective tools (risk scores and in this case, wich of them are used) or in subjective ways (clinical evaluation).

DETAILED DESCRIPTION:
This is an observational, cross-sectional, national multicenter study, trying to obtain local data about the global cardiovascular risk profile of patients attending ambulatory offices of general practitioners and cardiologists.

The aim of the study is to describe how physicians diagnose and stratify their patients in cardiovascular primary prevention setting and to highlight if patients are stratify through objective tools (risk scores and in this case, wich of them are used) or in subjective ways (clinical evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age, who give their written consent to take part.
* Patients without known vascular disease (primary prevention) under follow-up by the investigator, whose medical records have been initiated during the last 3 years.
* Patients who have completed their baseline CV risk assessment Lipid lowering treatment naive patients at the time of the stratification.

Exclusion Criteria:

* Incomplete or missing medical record data.
* Subjects with prior cardiovascular disease (peripheral vascular disease, coronary or cerebrovascular disease) symptomatic or asymptomatic.
* Subjects with terminal status disease or short life expectancy.
* Hypothyroidism without proper control.
* Pregnancy.
* Medical records compiled within a period longer than 3 years to the date of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, without known vascular disease (primary prevention) under follow-up by the investigator, whose medical records were initiated during the past 3 years and have completed their baseline assessment of CV risk
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Desciption of the assessment methods used to define the cardiovascular risk profile of patients attending outpatient medical consultation. | Day 1
  It will be evaluated the cardiovascular risk score for each patient. The proportion of use of each of the validated risk scores, as a tool of individual cardiovascular risk stratification and the proportion of use of a subjective assessment as tools of individual cardiovascular risk stratification used by general practitioners and cardiologists will be described.

SECONDARY OUTCOMES:
Comparison of the subjective individual risk assessment vs. the objective assessment obtained by the WHO risk score. | Day 1
  Comparison of the subjective individual risk assessment performed by the investigator for each patient at the moment of the risk stratification vs. the objective assessment obtained by the WHO risk score.
Comparison of the objective individual risk assessment achieved by the use of any risk score chosen by the treating physician in his / her usual practice vs. the objective assessment obtained by WHO risk score. | Day 1
  Comparison of the objective individual risk assessment achieved by the use of any risk score chosen by the treating physician in his / her usual practice for each patient at the moment of the risk stratification vs. the objective assessment obtained by WHO risk score.
Description of the treatment used, according to risk group and by the specialty of the treating physician. | Day 1
  Description of the pharmacological treatment implemented by the treating physician after risk stratification, according to cardiovascular risk group and by the specialty of the treating physician (cardiologists or GPs), such us Lipid Lowering drugs, antihypertensives, antiplatelet drugs, antidiabetic drugs.
Description of the extent of use of other diagnostic methods to define the individual cardiovascular risk (imaging scans, biomarkers). | Day 1
  Description of use of other diagnostic methods to define the individual cardiovascular risk, such us PCR, Apo A / Apo B, Homocysteine, Neck Vessels Ecodoppler, Echocardiogram, Ca Score, PEG, Ecostress - Gamma camera, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Buenos Aires, Argentina